CLINICAL TRIAL: NCT06493916
Title: Evaluation of Endotracheal Tube Cuff Pressure Measurements
Brief Title: Measurement of Endotracheal Tube Cuff
Status: Active, not recruiting | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Cevdet YARDIMCI, Asist. Prof. Dr., Bozok University
Other Study IDs: 2024-05-006
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Endotracheal Tube Cuff Pressure Levels in Practice
Keywords: Endotracheal tube cuff pressure; Endotracheal tube cuff pressure manometer; Endotracheal tube cuff pressure measuring; Manometer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endotracheal Intubated Group: Endotracheal tube insertion applied group

SUMMARY:
The purpose of this study is to evaluate whether the endotracheal intubation practitioners accordance to the literature knowledge of cuff pressure limits.

ELIGIBILITY:
Inclusion Criteria:

Intubated Patients

Exclusion Criteria:

No intubation Hemodynamically unstability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All intubated patients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-09-03 (Estimated); Study Completion 2024-10-03 (Estimated)

PRIMARY OUTCOMES:
Endotracheal tube cuff pressure measurements | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cevdet YARDIMCI, Principal Investigator — Anesthesiology and Reanimation
Locations (1):
- Yozgat Bozok Üniversitesi Araştırma ve Uygulama Hastanesi, Yozgat, Merkez/Yozgat, Turkey (Türkiye)